CLINICAL TRIAL: NCT04847583
Title: A Phase 2 Open-Label, Randomized Controlled Trial to Evaluate the Biomarker Change, Efficacy, Pharmacokinetics, Safety and Tolerability of Telacebec in Participants With Moderate COVID-19 Disease
Brief Title: A Phase 2 Study to Evaluate Biomarker Change, Efficacy, Pharmacokinetics, Safety and Tolerability of Telacebec (Q203) in Covid-19 Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q203-COVID-P2-ZA001
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-04

CONDITIONS: COVID-19 Virus Infection
MeSH Terms: conditions — COVID-19 | interventions — telacebec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telacebec (Q203) with COVID-19 standard of care (SoC) (Experimental)
  Interventions: Drug: Telacebec; Drug: COVID-19 Standard of care
- COVID-19 Standard of care (SoC) (Active Comparator)
  Interventions: Drug: COVID-19 Standard of care

INTERVENTIONS:
Drug: Telacebec — Telacebec 100 mg tablet
  Other Names: Q203
  Arms: Telacebec (Q203) with COVID-19 standard of care (SoC)
Drug: COVID-19 Standard of care — The Standard of Care treatment and administration thereof will be determined by the Investigator

SUMMARY:
This is a Phase 2, open-label, randomized controlled trial to determine the effects of Telacebec (Q203) on inhibition of leukotriene production, clinical change, pharmacokinetics, and safety in participants with moderate COVID-19 disease

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all study-related procedures.
2. Provide written, informed consent to undergo Human Immunodeficiency Virus (HIV) testing.
3. Willingness and ability to attend scheduled visits and undergo study assessments.
4. Able and willing to measure their oxygen saturation level and temperature, record their COVID-19 symptoms and complete a patient diary.
5. Male or female aged 18 years or older.
6. Confirmed and documented SARS-CoV-2 infection, defined as RT-PCR laboratory confirmation.
7. Clinical and/or radiological findings indicative of moderate COVID-19 disease

Exclusion Criteria:

1. Severe or critical COVID-19 disease at enrollment (Day 1) (per NIH Treatment Guideline categorization) as determined by the Investigator.
2. Inability to swallow oral medication.
3. Concurrent known asthma, active tuberculosis or tuberculosis within the last 3 months, or any other condition that could compromise the well-being of the participant, or prevent, limit or confound protocol specified assessments, in the opinion of the Investigator.
4. Female Participant who is pregnant, breast-feeding, or planning to conceive a child within the anticipated period of participating in the study or within 6 months after last dose of study medication. Males planning to conceive a child during the study or within 6 months of cessation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Biomarker change | Day 1 and 14
  Percentage Inhibition of whole blood Leukotriene B4 (LTB4) production at 4 hours post dose SoC versus SoC plus telacebec

CONTACTS AND LOCATIONS:
Locations (3):
- South Africa (3):
  - Chris Hani Baragwanath Academic Hospital, Soweto, Gauteng
  - KwaPhila Health Solutions, Durban, Kwa-Zula Natal
  - TASK Eden, George, Western Cape

IPD SHARING:
Plan to Share IPD: Undecided